CLINICAL TRIAL: NCT03898999
Title: Relationship of the Ankle ROM With Balance and Falls in Older Adults: Observational Study
Brief Title: Relationship of de Ankle ROM With Balance and Falls in Older Adults
Acronym: ANKLE_JOINT
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández, Principal Investigator, University of Valencia
Other Study IDs: DHG04
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Aging Problems
Keywords: Ankle; Balance; Falls; Older Adult
MeSH Terms: interventions — Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adult: Individuals belonging to the population group of the elderly (60 years or more)
  Interventions: Other: Overall status

INTERVENTIONS:
Other: Overall status — An assessment is made of the participants measuring both the joint range of the ankle and the balance and risk of falls.

SUMMARY:
The ankle is an important joint to maintain a good balance within the population of the older adult. As people get older, problems appear in this joint. Many of these problems affect the correct joint range of the ankle. There is evidence to suggest that a lower range of motion in the ankle can negatively affect balance and, consequently, increase the risk of falls in the elderly. It would be interesting to assess if this relationship is true. The aim of the study will be to study if the state of the joint range of the ankle is related in some way to balance and falls in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older

Exclusion Criteria:

* Do not sign the informed consent
* Lower limb injury in the previous three months
* Presenting severe pathology that affects balance or mobility

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects must belong to the population of older adults, who must not present serious pathologies that make their balance or mobility difficult, although they can use aids.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Lunge Test (°) | Baseline
  Measure of weight-bearing ankle dorsiflexion with an inclinometer.
Active Ankle Range of Movement | Baseline
  Measure of the active range of movement of the ankle with a telescopic goniometer.

SECONDARY OUTCOMES:
Pressure Platform - Open Eyes | Baseline
  Measure static balance. Quantitative assess of area and speed of swing, with open eyes.
Pressure Platform - Closed Eyes | Baseline
  Measure static balance. Quantitative assess of area and speed of swing, with closed eyes.
One Leg Balance | Baseline
  Measure balance ability to maintain in monopodal stance, towards registering time.
Timed "Up and Go" Test | Baseline
  Measures the functional mobility and dynamic balance, through a circuit where the subject will have to get up, walk and sit down.
Functional Reach | Baseline
  Measure the limits of stability, calculating the distance that can move the center of gravity forward without falling.
Falls Efficacy Scale-International | Baseline
  Is a scale that, through 16 items, describes the concern that a subject has to suffer a fall.
Register of falls | Baseline
  The number of falls that the subject has suffered in the last year is collected.
Ankle plantar flexion strength | Baseline
  The plantar flexion strength is measured by means of a dynamometer, is related with the risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, Principal Investigator — University of Valencia; Jose M Blasco, PhD, PT, Study Director — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided